CLINICAL TRIAL: NCT05796804
Title: Erector Spinae Block Versus PENG Block for Postoperative Analgesia After Total Hip Replacement
Brief Title: Erector Spinae Block Versus PENG Block for Hip Replacement
Acronym: PENGESP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Papa Giovanni XXIII Hospital (Other)
Responsible Party: Principal Investigator, Dario Bugada, MD, Papa Giovanni XXIII Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 030/23
Record Dates: First submitted 2023-03-21; First posted 2023-04-04 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERECTOR SPINAE PLANE BLOCK (Active Comparator): ultrasound guided block at L4
  Interventions: Procedure: ERECTOR SPINAE PLANE BLOCK; Procedure: spinal anesthesia
- PERICAPSULARE NERVE GROUP AND LATERAL FEMORAL CUTANEOUS NERVE BLOCK (Active Comparator): ultrasound guided block below the ileo-psoas muscle tendon, above the ilio-pectineous eminence and ultrasound guided block of lateral femoral cutaneous nerve
  Interventions: Procedure: Peng block + lateral femoral cutaneous nerve block; Procedure: spinal anesthesia

INTERVENTIONS:
Procedure: ERECTOR SPINAE PLANE BLOCK — ULTRASOUND GUIDED - ROPIVACAINE 30 ml 0.5%
  Arms: ERECTOR SPINAE PLANE BLOCK
Procedure: Peng block + lateral femoral cutaneous nerve block — ULTRASOUND GUIDED - ROPIVACAINE 20 ml 0.5% + 10 ml 0.5%
  Arms: PERICAPSULARE NERVE GROUP AND LATERAL FEMORAL CUTANEOUS NERVE BLOCK
Procedure: spinal anesthesia — bupivacaine 0.5% 2.2 ml

SUMMARY:
THR (Total Hip Replacement) can be very painful and regional anesthesia is very effective in reducing postoperative pain. Erector Spinae Plane Block (ESPB) and PENG (pericapsular nerve group block) are alternative approaches to the hip sensitive nerve branches that resulted to be very promising for hip surgeries. However, no studies investigated the analgesic superiority of either PENG or ESPB. In our study the investigators compare PENG (with a lateral femoral cutaneous nerve block) and ESPB in terms of pain relief expressed as morphine consumption in the first 24 hours after primary THR.

ELIGIBILITY:
Inclusion Criteria:

* primary total hip replacement
* informed consent

Exclusion Criteria:

* allergies to study drugs
* spinal anesthesia contraindicated
* kidney failure
* epilepsy, psychiatric disease, neurologic deficits
* revision surgery
* neuropathies in the lumbar area
* no informed consent
* pregnancy
* alcohol/opioid abuse
* emergency surgery/intensive care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-04-13 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
morphine consumption | 24 hours
  milligrams of morphine by patient controlled analgesia intravenously

SECONDARY OUTCOMES:
postoperative pain | 48 hours
  numeric rating scale - NRS 11 point scale from 0 = "no pain" to 10 = "worst imaginable pain"
neuropathic pain | 48 hours
  DN4 questionnaire - 4 items questionnaire to investigate the occurrence of neuropathic component
postoperative complications | 48 hours
  nausea, vomiting, vertigo, blurred vision, syncope, bleeding, falls
chronic postoperative pain | 3 months
  numeric rating scale 11 point scale from 0 = "no pain" to 10 = "worst imaginable pain"

CONTACTS AND LOCATIONS:
Locations (1):
- Aast Papa Giovanni Xxiii, Bergamo, Italy

IPD SHARING:
Plan to Share IPD: No